CLINICAL TRIAL: NCT03850951
Title: Assessment of Dentoalveolar Changes Resulting From Orthodontic Treatment of Crowding With Fixed Lingual Orthodontic Appliances Versus Fixed Labial Orthodontic Appliances. 'A Clinical Randomized Controlled Trial
Brief Title: Comparison Between Lingual and Labial Fixed Orthodontic Appliances in the Treatment of Crowding Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-04-2018
Record Dates: First submitted 2018-12-17; First posted 2019-02-22 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Crowding
Keywords: Fixed appliances; labial appliances; lingual appliances
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lingual appliances "AO®" (Experimental): Patients with moderate crowding will be treated without extraction using lingual fixed appliances from American Orthodontics company.
  Interventions: Device: Lingual appliances
- Labial appliances "AO®" (Experimental): Patients with moderate crowding will be treated without extraction using labial fixed appliances from American Orthodontics company.
  Interventions: Device: Labial appliances

INTERVENTIONS:
Device: Lingual appliances — Patients with moderate crowding will be treated without extraction using lingual appliances.
  Arms: Lingual appliances "AO®"
Device: Labial appliances — Patients with moderate crowding will be treated without extraction using labial appliances.
  Arms: Labial appliances "AO®"

SUMMARY:
Patients who have moderate crowding that could be treated without extraction will be treated in this study using either lingual or labial fixed orthodontic appliances. All patients will receive a cone-beam computed tomography (CBCT) scan in two different times (T0: before treatment, T1: after treatment). The dentoalveolar changes will be assessed.

DETAILED DESCRIPTION:
Lingual orthodontic appliances provide an ultimate esthetic solution for patients who do not want visible orthodontic appliances. Recently, lingual orthodontic treatment outcomes have become similar and comparable to those produced with labial orthodontic treatment. However, placement of orthodontic brackets on the lingual surfaces of teeth causes changes in their morphology, which results in articulation problems, chewing difficulties, tongue irritation and other impairments. In this respect, the main difference between the labial and lingual techniques is the distance between the point of application of the force that is transmitted through the bracket and the centre of resistance of the tooth. Consequently, the displacement and stress induced in bone by these two techniques will also differ, and these need to be evaluated so that useful comparisons can be made between these two techniques. Patients who have moderate crowding that could be treated without extraction will be treated in this study using either lingual or labial fixed orthodontic appliances. All patients will receive a cone-beam computed tomography (CBCT) scan in two different times (T0: before treatment, T1: after treatment). The dentoalveolar changes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Class I malocclusion.
* Moderate crowding in the dental arch (3 to 5-mm tooth-size arch-length discrepancy).

Exclusion Criteria:

* Inappropriate oral hygiene and periodontal diseases.
* Previous orthodontic treatment.
* Craniofacial syndromes, cleft lip and/or palate (soft and/or hard).
* Subject with systemic diseases.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Dentoalveolar changes after crowding treatment | Changes will be evaluated before and after crowding treatment which will take approximately 12 months
  Dentoalveolar changes before and after crowding treatment will be evaluated using CBCT.

SECONDARY OUTCOMES:
ABO- Objective Grading System | After treatment completion, an average of 1 year
  Objective grading system phase III examination will be done to systematically grade post treatment records. The ABO-OGS contains eight criteria: alignment, marginal ridges, buccolingual inclination, occlusal relationships, occlusal contacts, overjet, interproximal contacts and root angulation. Patients will be deducted for any discrepancy from ideal as described by the ABO. Every case that loses 30 or fewer points generally receives a passing grade for the ABO phase III examination.
Change in oral health related quality of life | (1) at the beginning of the treatment, (2) after week, (3) after 2 weeks, (4) after 4 weeks, (5) after 6 months, (6) after treatment completion, an average of 1 year.
  Patients in both groups will be given a questionnaire to be filled. The questionnaire to be used is called Oral-Health-Impact-Profile with 14 items (OHIP-14) which can be filled in 3 minutes. OHIP-14 includes a subjective evaluation of the individual's oral health, functional well being, emotional well being, expectations and satisfaction with care and sense of self.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S Burhan, PhD., Study Director — Faculty of Dentistry, Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The Individual participant data will be only available for the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Background] Fritz U, Diedrich P, Wiechmann D. Lingual technique--patients' characteristics, motivation and acceptance. Interpretation of a retrospective survey. J Orofac Orthop. 2002 May;63(3):227-33. doi: 10.1007/s00056-002-0124-3. English, German. PMID 12132310
- [Background] Jacobs C, Gebhardt PF, Jacobs V, Hechtner M, Meila D, Wehrbein H. Root resorption, treatment time and extraction rate during orthodontic treatment with self-ligating and conventional brackets. Head Face Med. 2014 Jan 23;10:2. doi: 10.1186/1746-160X-10-2. PMID 24456620
- [Background] Khattab TZ, Farah H, Al-Sabbagh R, Hajeer MY, Haj-Hamed Y. Speech performance and oral impairments with lingual and labial orthodontic appliances in the first stage of fixed treatment. Angle Orthod. 2013 May;83(3):519-26. doi: 10.2319/073112-619.1. Epub 2012 Oct 18. PMID 23075062
- [Background] Klang E, Beyling F, Knosel M, Wiechmann D. Quality of occlusal outcome following space closure in cases of lower second premolar aplasia using lingual orthodontic molar mesialization without maxillary counterbalancing extraction. Head Face Med. 2018 Sep 24;14(1):17. doi: 10.1186/s13005-018-0176-2. PMID 30249268
- [Background] Pauls AH. Therapeutic accuracy of individualized brackets in lingual orthodontics. J Orofac Orthop. 2010 Sep;71(5):348-61. doi: 10.1007/s00056-010-1027-3. Epub 2010 Oct 21. English, German. PMID 20963544
- [Background] Pauwels R. Cone beam CT for dental and maxillofacial imaging: dose matters. Radiat Prot Dosimetry. 2015 Jul;165(1-4):156-61. doi: 10.1093/rpd/ncv057. Epub 2015 Mar 23. PMID 25805884
- [Background] Tian YL, Liu F, Sun HJ, Lv P, Cao YM, Yu M, Yue Y. Alveolar bone thickness around maxillary central incisors of different inclination assessed with cone-beam computed tomography. Korean J Orthod. 2015 Sep;45(5):245-52. doi: 10.4041/kjod.2015.45.5.245. Epub 2015 Sep 23. PMID 26445719